CLINICAL TRIAL: NCT06890949
Title: Evaluation Of Occlusal Wear Of Bioflx Crowns Compared To Zirconia Crowns On Primary Molars
Brief Title: Occlusal Wear Of Bioflx Crowns Compared To Zirconia Crowns On Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eithar Musa Abdelrahman Hussien, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OW-BFC VS ZRC
Record Dates: First submitted 2025-03-15; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Carious Primary Molars

STUDY DESIGN:
Who Masked: Participant
Masking Description: statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- (Group A : preformed Bioflx crown (Experimental): Kids-e-Dental LLP (ANDHERI, MUMBAI, INDIA) introduced Bioflx Crowns and claimed as the first flexible, durable, and esthetic preformed crown for primary molars. Bioflx Crowns are monochromatic, metal-free, tooth-colored crowns made up of high- strength resin polymer used in the medical device industry having high strength, flexibility, and durability. These crowns are autoclavable and are like SSC in tooth preparation as claimed by the manufacturer. Their flexibility and snap-fit technology aim to improve retention while minimizing trauma during placement
  Interventions: Other: (Group A: Preformed Bioflx Crown)
- (Group B: Preformed zirconia crown) (Experimental): NuSmile Zirconia Crowns are prefabricated, esthetic full-coverage restorations designed for primary teeth. Known for their superior strength, durability, and natural tooth-like appearance, these crowns provide an excellent alternative to traditional stainless steel crowns. Made from high-quality medical-grade zirconia, they are biocompatible, resistant to chipping, and highly polished to minimize plaque accumulation and gingival irritation.
  NuSmile Zirconia Crowns require significant tooth preparation for proper fit and retention. They are available in various sizes to accommodate different primary molars and anterior teeth. Their lifelike translucency and color-matching capabilities make them a preferred choice for parents and clinicians seeking a highly esthetic and long-lasting pediatric restoration
  Interventions: Other: (Group B: Preformed Zirconia crown)

INTERVENTIONS:
Other: (Group A: Preformed Bioflx Crown) — Crown Selection & Tooth Preparation
  Measure the mesiodistal width using calipers to select an appropriately sized crown.
  If a mesial or distal wall is missing, use the contralateral tooth for size selection.
  Choose the crown that closely matches the measured mesiodistal width. Select the smallest crown that preserves proximal contacts using a trial-and-error approach.
  if crimping is necessary use Howe's pliers.
  Tooth Preparation Perform 1-1.5 mm occlusal reduction using a tapered diamond bur. Reduce proximal areas by approximately 0.5 mm to clear the contact area.
  Crown Placement & Cementation Ensure a snug fit of the selected crown. Apply a thin layer of glass ionomer cement inside the crown. Seat the crown firmly using finger pressure. Have the child bite down gently to ensure proper seating.
  Final Adjustments & Cleanup Remove excess cement with floss or an explorer. Verify the crown's fit, occlusion, and stability.
  Arms: (Group A : preformed Bioflx crown
Other: (Group B: Preformed Zirconia crown) — Crown Selection
  Measure the mesiodistal width using calipers to select the appropriate crown. If a mesial or distal wall is missing, use the contralateral tooth for size selection.
  Choose the crown that closely matches the measured width. Select the smallest crown that preserves proximal contacts.
  Tooth Preparation
  Reduce the occlusal surface by 1.5-2 mm using a tapered diamond bur. Reduce interproximal areas by 1-1.5 mm, ensuring a feather-edge finish. Perform a 1-2 mm subgingival preparation using a tapered fissure bur.
  Crown Placement & Passive Fit Check
  Place the selected crown and check for passive fit.
  Cementation of the Crown
  Apply a thin layer of glass ionomer cement inside the crown. Seat the crown with passive finger pressure. Have the child bite down gently to ensure proper seating.
  Final Adjustments & Cleanup
  Remove excess cement using floss or an explorer. Verify fit, occlusion, and stability
  Arms: (Group B: Preformed zirconia crown)

SUMMARY:
The goal of this clinical trial is to evaluate the occlusal wear of Bioflx crowns compared to zirconia crowns in the restoration of primary molars.

The main question[s] it aims to answer : " Is there a difference in the occlusal wear of BioFlx crowns compared to zirconia crowns in the restoration of primary molars?" The study will also assess the clinical performance of both types of crowns in terms of retention,gingival health, preparation time, as well as child and parental satisfaction.

DETAILED DESCRIPTION:
Occlusal wear is a critical factor in determining the longevity and functional efficiency of dental restorations, especially in pediatric patients. Primary molars undergo significant masticatory forces, which can lead to material wear and affect the restoration's durability. Bioflex (a relatively new material) and zirconia crowns are commonly used for full-coverage restorations in primary molars, yet there is limited research comparing their occlusal wear characteristics. Understanding how these materials perform under occlusal forces can guide clinicians in selecting the most suitable material for pediatric dental restorations Dental caries in primary molars represent a significant issue within pediatric dentistry. In cases where traditional fillings prove insufficient, full coronal coverage becomes necessary. Stainless steel crowns (SSCs) have long been the standard due to their durability and cost-effectiveness, but their metallic appearance has led to increased interest in aesthetic alternatives like zirconia and Bioflx crowns.

Zirconia offers improved aesthetics, biocompatibility, and mechanical strength, though its long-term clinical performance remains underexplored. While zirconia crowns provide durability and superior aesthetics, they require significant tooth preparation, which may compromise tooth structure. Bioflx crowns, a newer option, combine the benefits of stainless steel and zirconia with more flexibility and less tooth reduction. However, comparative studies on their clinical efficacy, occlusal wear, and patient satisfaction are still needed.

Zirconia offers improved biocompatibility, mechanical strength, and enhanced esthetics, but limited comparative data exists regarding its clinical performance.

The growing awareness among parents regarding the importance of maintaining primary teeth until their natural shedding necessitates a thorough evaluation of the durability, wear resistance, retention, gingival response, and overall clinical efficacy of these crown materials. Zirconia crowns have been the preferred choice for aesthetic restorations due to their natural appearance and durability. However, their requirement for excessive tooth preparation poses challenges in pediatric patients.

Bioflx crowns, made from a biocompatible hybrid resin polymer, offer a flexible fit with minimal tooth reduction while maintaining aesthetic appeal. A comprehensive comparison of occlusal wear between these two materials is crucial for assisting clinicians in selecting the most suitable restorative solution for primary molars. This research seeks to offer evidence-based guidance by evaluating the long-term clinical performance of Bioflx crowns in relation to zirconia crowns.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 4 and 8 years with primary molar that needs to be covered by crown.
2. Medically healthy children (ASA I or II according to the American Society of Anesthesiologists classification).
3. Children whose parent or guardian are willing to sign an informed consent.
4. Children whose parent or guardian are willing to comply with follow-up visits. -
5. Frankl's positive and definitely positive patient

Exclusion Criteria:

1. Molars with severe structural loss that may compromise crown retention.
2. Children with poor oral hygiene that may contribute to higher plaque levels and affect the clinical outcomes of the crown restorations.
3. Children with history of allergies; Known allergies to dental local anesthesia or to the materials used in Bioflx crowns.
4. Children with any systemic conditions or disabilities that may affect their ability to participate in the study.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Occlusal wear of crown | T (Time): 12months interval T0: 0 T1: 3 month T2: 6month T3: 12 month]
  Measure by Modified United States Public Health System criteria:
  Alpha: Occlusal surface intact. Bravo: Wear of occlusal surface without tooth surface exposure Charlie: Wear of occlusal surface with exposure

SECONDARY OUTCOMES:
Retention | [Time Frame: follow-up:T (Time): 12months interval T0: 0 T1: 3month T2: 6month T3 : 12 month]
  Measure by :Modified United States Public Health System criteria:Alpha: Intact Bravo:Chipped/loss of material Charlie: Complete loss of crown
Gingival Health | T (Time): 12 months interval T0: 0 T1: 3month T2: 6month T3 : 12 month]
  Measure by: Gingival index:
  0: healthy gum
  1. mild discoloration and edematous gingiva no bleeding on probing
  2. red oedematous and shiny gingiva bleeding on probing
  3. red oedematous and ulceration gingiva spontaneous bleeding
preparation time | [Time Frame: baseline]
  Measure by : Stopwatch per minutes.
child and parental satisfaction | [Time Frame: T (Time): 12months interval T0: 0 T1: 3 month T2: 6month T3: 12 month]
  Measure by: 5-Point likert's scale units of measurement
  1. very happy
  2. happy
  3. neither
  4. unhappy
  5. very unhappy / Questionnaire:Ordinary or N/ A existing validated tool

CONTACTS AND LOCATIONS:
Overall Officials: Manal Ahmed Elshiekh, prof, PhD, Study Director — Cairo University
Locations (1):
- Faculty of dentistry cairo university, Cairo ,Giza, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahate I, Fulzele P, Thosar N. Comparative evaluation of clinical performance, child and parental satisfaction of Bioflx, zirconia and stainless steel crowns in pediatric patients. F1000Res. 2023 Dec 21;12:756. doi: 10.12688/f1000research.133464.2. eCollection 2023. PMID 38911945